CLINICAL TRIAL: NCT01063777
Title: Exercise Therapy and Patient Education for Individuals With Hip Osteoarthritis. Long-term Follow-up of a Prospective, Randomized Controlled Intervention Study.
Brief Title: Exercise Therapy and Patient Education for Individuals With Hip Osteoarthritis. Long-term Follow-up.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Sponsor
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03c-2009-NAR
Record Dates: First submitted 2010-02-04; First posted 2010-02-05 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Osteoarthritis, Exercise therapy, Patient Education
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Patient Education as Topic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Other: A 12 week exercise therapy program and patient education.
- 2 (Active Comparator)
  Interventions: Other: Patient education

INTERVENTIONS:
Other: A 12 week exercise therapy program and patient education. — The exercise protocol includes exercises from former studies on comparable patient populations. The intensity of the strength- and flexibility exercises meets the American College of Sports Medicine's (ACSM) recommendations for developing and maintaining muscular fitness in adults.Patients will be required to exercise for 60 minutes, three days a week for 12 weeks. Patient's attendance to the exercise program (compliance) will be registered by the physical therapists.
  All patients included in the study will receive two individual and three small-group (6-7 patients) sessions lasting one hour each time.
  Arms: 1
Other: Patient education — All patients included in the study will receive two individual and three small-group (6-7 patients) sessions lasting one hour each time.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the long term effect of exercise therapy and patient education compared to patient education only in individuals with hip OA, and to evaluate predictive factors for changes in hip osteoarthritis both clinically and on x-ray.

Main hypothesis H01: There are no significant long term ( 2 years) differences in hip function, quality of life, physical function and radiological changes between those individuals who went through a patient education program and a 12 week exercise therapy program compared to patient education program only.

Material and Methods:

109 patients with radiographically verified hip OA are included in the randomized controlled trial; randomized to 12 week exercise therapy program and patient education (n=55) and patient education program only (n=54).

Data will be collected 2 years after completed intervention period in the original RCT, and 6 months and 2 years postoperatively for those patients who have undergone total hip arthroplasty.

The main outcome is:

The Disease Specific WOMAC-Index.

Secondary outcome measures are:

Hip X-ray, SF-36v2 (quality of life),PASE (activity score), Self-efficacy for pain, isokinetic muscle strength tests, 6 minute walk test, Åstrand's bike test, range of motion.

Status:

This study is a prolongation of an on-going RCT (3a-2005-NAR). The inclusion, intervention and follow-ups including 1 year follow-up is completed. 2 year post-intervention follow-up will be completed in 2010, 2 year follow-up postoperative for patients undergoing total hip artroplasty will continue throughout 2011.

The study will be carried out: NAR-Orthopedic Centre, Ullevaal University Hospital.

DETAILED DESCRIPTION:
Aims

Aim 1 To evaluate the long-term effects of a patient education program and a 12 week exercise therapy program (IG) compared to patient education only (CG) on hip function, quality of life and physical function in patients with hip OA not eligible for total hip arthroplasty (THA) at time of inclusion Aim 2

1. To examine differences in radiographic changes between those individuals who went through a patient education program and a 12 week exercise therapy program (IG) compared to those who only went through a patient education program (CG) 2 years after inclusion.
2. To examine predictive factors for radiographic changes and changes in hip function at a 2 year follow-up after inclusion.

Aim 3

1. To evaluate hip function, quality of life and physical function in those patients who have gone through total hip arthroplasty (THA)
2. To examine differences in hip function, quality of life, and physical function in patients who prior to surgery went through a patient education program and a 12 week exercise therapy program (IG) compared those patients who went through a patient education program only (CG) 6 months after THA.

Material and methods

Design:

This study is a prospective, randomized clinical trial examining the long term effect of two different interventions for patients with hip OA. The long term follow-up is based on an ongoing study (03a-2005-NAR) on short term outcome.

Patients:

109 patients were recruited from Orthopaedic Center, Ullevål University Hospital, NIMI, and Diakonhjemmet Hospital, Oslo from April 2005 till October 2007.

Inclusion Criteria:

Patients between 40 and 80 years old with uni- or bilateral hip disability not eligible for hip surgery will be recruited from Orthopaedic Centre, Ullevål University Hospital, NIMI, and Diakonhjemmets Sykehus (Hospital), Oslo. Inclusion criteria for all subjects are:

* Harris Hip Score (35) between 60 and 95, and hip pain of more than 3 months.
* Radiographic verified hip OA,classified by an orthopaedic surgeon (LN), according to Danielsson's criteria for radiographic hip OA.

Exclusion Criteria:

Patients will be excluded if they have a history of resent trauma or functional impairment to the lower limbs or diseases which might interfere with participation (rheumatoid arthritis, cancer, osteoporosis, severe back pain, knee OA).

Patients with co-morbidities not tolerating physical activities will be excluded.

Interventions:

The interventions are described in the registration concerning the short-term follow-up study (03a-2005-NAR).

Outcome Measurements:

The primary end point for Aim 1 and 3 is WOMAC (hip function), and the primary endpoint for Aim 2 is radiographic changes using the Danielsson's criteria for minimal joint space.

Pain and Functional Activity: The primary (main) outcome measurement is the self-reported functional outcome measure, the disease-specific questionnaire Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). WOMAC is found to be a valid, reliable and responsive outcome measure in patients with hip OA.

The self-reported Physical Activity Score for the Elderly (PASE) will be used to record the individuals activity level prior to inclusion and at follow-up intervals. Hip pain will be recorded on a visual analogue scale (VAS) rating from 0 to 100 mm; 0 represents "no pain" and 100 represents "as much pain he/she can possibly imagine". The pain will be recorded after the 6 minutes walking test (se below).

Six minute walk test (Enright, 2003): Observed functional capacity and cardiovascular fitness will be assessed by a six minute walk test. This test has been reliability estimated for older adults and validated for older adults and individuals with total hip arthroplasty.

Health related quality of life and pain management: Quality of life will be assessed by using the self-administered generic questionnaire 36-item short-form health survey (SF-36) version 2.

Muscle strength: Isokinetic muscle strength will be tested in Technogym REV 9000 (Gambettola, Italia) and measured as peak torque at 60°s-1 for hip flexion/extension, knee flexion/extension and ankle flexion/extension.

Cardiovascular Fitness (Åstrand & Rodahl, 1986): Tested by a sub-maximal bicycle ergometer test according to the method described by Åstrand & Rodahl. The load will be adjusted to each subject. Results will be corrected for age and gender and expressed in ml O2 / kg / min.

Range of motion: Measured with a plastic goniometer. Flexion, abduction, and adduction is registered in supine position, with a fixation of the contralateral leg. Internal and external rotation is registered in prone position with fixation over buttocks. Extension is registered according to Thomas test.

Radiographic examination: Hip X-rays will be taken at inclusion and at 2 year follow-up, and are classified by an orthopaedic surgeon (LN), according to Danielsson's criteria for radiographic hip OA.

Data Collections and Follow-Up:

Data will be collected at inclusion, after the 12 weeks intervention period, and at follow-ups at 6 months, 1 year and 2 years. Data from all outcome measurements will be collected from all patients at all follow-ups, except at 1 year follow-up, where only the questionnaires will be included. Radiographic examination is only included at inclusion and at 2 year follow-up.

Power Calculations:

The WOMAC Index is the main outcome measurement. Power calculations based on a standard deviation of 23 mm, and a minimum clinically important difference of 15 mm between groups calculated that there is a need for 49 patients in each group. To account for drop-outs, a total of 109 patients is included in the RCT.

Blinding:

Personnel responsible for the intervention will not be involved in data collection. Physical therapists collecting data will be blinded for patients' group allocation. A research coordinate person, not involved in any part of the study intervention or data collections, will be responsible for randomization procedures (give subjects information about group allocation)

Statistical Analysis:

Data in the randomized controlled trial will be analyzed both according to the intention to treat principles and additional analysis for the compliers adhering to the exercise protocol at a cut-off value of 24 or more training sessions.

Registration of Complications, Drop-Outs and Compliance:

Complications and drop-outs will be registered by persons responsible for data collection. There will be used intention to treat analysis. Compliance to the patient education and the exercise protocol will be registered by the physical therapists responsible for the treatment.

Ethics:

All patients and control subjects will receive written and oral information about the study and sign an informed consent before inclusion. The project will be performed according to recommendations of the Helsinki Declaration. Approval is obtained from the Regional Committee of Medical Research Ethics.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 80 years old with uni- or bilateral hip disability
* Harris Hip Score (36) between 60 and 95. Harris Hip score (0-100 points) is widely used as an assessment of hip function in patients with hip OA. Harris Hip Score of 60 or below are used regularly at our institution as one of the criteria for hip surgery (arthroplasty).
* Patients will be included if they have more than 3 months of hip pain.
* Patients with radiographic verified hip OA (Danielson's criteria for radiographic OA: Danielsson's criteria for minimal joint space: < 4 mm < 70 years, < 3 mm ≥ 70 years, or 1 mm difference between hips).

Exclusion Criteria:

* Patients have a history of resent trauma or functional impairment to the lower limbs or diseases which might interfere with participation (rheumatoid arthritis, cancer, osteoporosis, severe back pain, knee OA).
* Patients with co-morbidities not tolerating physical activities

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 12 weeks, 6, 12 and 24 months.

SECONDARY OUTCOMES:
SF-36 (quality of life) | Baseline, 12 weeks, 6, 12 and 24 months.
PASE (activity score) | Baseline, 12 weeks, 6, 12 and 24 months.
Self-efficacy for pain | Baseline, 12 weeks, 6, 12 and 24 months.
Muscle strength tests | Baseline, 12 weeks, 6 and 24 months.
6 minute walk test | Baseline, 12 weeks, 6 and 24 months.
Åstrand's bike test | Baseline, 12 weeks, 6 and 24 months.
Range of motion | Baseline, 12 weeks, 6 and 24 months.
Radiographic examination | Baseline and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PT, PhD, Principal Investigator — NAR- Orthopedic Centre, Ullevål University Hospital
Locations (1):
- NAR-Orthopedic Centre, Ullevål University Hospital & Hjelp24 NIMI, Oslo, Norway

REFERENCES:
- See also: Homepage NAR — http://www.active-rehab.no